CLINICAL TRIAL: NCT04250714
Title: POLARx Cardiac Cryoablation System Post Market Clinical Follow-up Study
Brief Title: POLARx Cardiac Cryoablation System Study
Acronym: POLAR ICE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PY003
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Treatment patients: Subjects indicated for the treatment of AF with the cryoablation system according to current and future Guidelines and system indications for use
  Interventions: Device: Boston Scientific Cardiac Cryoablation System

INTERVENTIONS:
Device: Boston Scientific Cardiac Cryoablation System — cryoablation of atrial fibrillation consisting in electrical isolation of the pulmonary veins

SUMMARY:
This is a Post Market Clinical Follow-up (PMCF) study designed to establish the continued safety and effectiveness profile of the Boston Scientific Cardiac Cryoablation System after receiving CE mark.

DETAILED DESCRIPTION:
The study will provide information on real-world usage of the Boston Scientific Cardiac Cryoablation System when used to perform pulmonary vein isolation (PVI) for the ablation treatment of atrial fibrillation (AF), according to the current and future guidelines and product indications for use. This may include but not limited to: repeated ablations to treat AF, concomitant or delayed adjunctive ablation strategies with other products and use of different diagnostic products to validate the results such as 3D mapping systems.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects indicated for the treatment of AF with the cryoablation system according to current and future Guidelines and system indications for use;
2. Subjects who are willing and capable of providing informed consent;
3. Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center;
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Any known contraindication to an AF ablation or anticoagulation, including those listed in the instructions for use;
2. Subjects with indication for treatment of AF that is not according to current and future Guidelines and system indications for use;
3. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause;
4. Known or pre-existing severe Pulmonary Vein Stenosis;
5. Evidence of myxoma, LA thrombus or intracardiac mural thrombus;
6. Previous cardiac surgery (e.g. ventriculotomy or atriotomy, CABG, PTCA, stent procedure) within 90 days prior to enrollment;
7. Implantable cardiac device procedures (e.g. PM, ICD, CRT) within 30 days prior to enrollment;
8. Implanted Left Atrial Appendage Closure device prior to the index procedure;
9. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder;
10. Subjects with severe valvular disease OR with a prosthetic - mechanical or biological - heart valve (not including valve repair and annular rings);
11. Presence of any pulmonary vein stents;
12. Active systemic infection;
13. Vena cava embolic protection filter devices and/ or known femoral thrombus;
14. Any previous history of cryoglobulinemia;
15. History of blood clotting or bleeding disease;
16. Any prior history of documented cerebral infarct, TIA or systemic embolism (excluding a post-operative deep vein thrombosis (DVT)) ≤ 180 days prior to enrollment;
17. Subjects who are hemodynamically unstable;
18. The subject is unable or not willing to complete follow-up visits and examination for the duration of the study;
19. Life expectancy ≤ 1 year per investigator's opinion;
20. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon investigator's discretion);
21. Unrecovered/unresolved Adverse Events from any previous invasive Procedure;
22. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients indicated for the treatment of AF with isolation of pulmonary veins technique according to current and future Guidelines and system indications for use
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- UZ Brussel, Brussels, Belgium
- Klinicki Bolnicki Centar, Split, Croatia
- France (5):
  - CHU De Brest - Hopital de la Cavale Blanche, Brest
  - CHU De Caen, Caen
  - CHU Grenoble - Hopital Michallon, Grenoble
  - Clinique Pasteur, Toulouse
  - CHRU Hospital Trousseau, Tours
- Germany (4):
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Vivantes Klinikum Am Urban, Berlin
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
- Italy (3):
  - Maria Cecilia Hospital SPA, Cotignola
  - Centro Cardiologico Monzino, Milan
  - Ospedale S.G. Calibita Fatebenefratelli - Isola Tiberina, Roma
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Isala Klinieken, Zwolle
- United Kingdom (3):
  - Papworth Hospital, Cambridge
  - Liverpool Heart and Chest Hospital, Liverpool
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Luik A, Anic A, Martin CA, Tilz RR, Yap SC, de Asmundis C, Champ-Rigot L, Iacopino S, Sommer P, Albrecht EM, Raybuck JD, Richards E, Cielen N, Defaye P. One-Year Success Rates of a Stable, Low Pressure Cryoballoon for the Treatment of Paroxysmal Atrial Fibrillation: Results of the Prospective, International, Multicenter POLAR ICE Study. J Cardiovasc Electrophysiol. 2025 May;36(5):1046-1052. doi: 10.1111/jce.16645. Epub 2025 Mar 19. PMID 40108686
- [Result] Martin CA, Tilz RRR, Anic A, Defaye P, Luik A, de Asmundis C, Champ-Rigot L, Iacopino S, Sommer P, Albrecht EM, Raybuck JD, Richards E, Cielen N, Yap SC; POLAR ICE Investigators. Acute procedural efficacy and safety of a novel cryoballoon for the treatment of paroxysmal atrial fibrillation: Results from the POLAR ICE study. J Cardiovasc Electrophysiol. 2023 Apr;34(4):833-840. doi: 10.1111/jce.15861. Epub 2023 Feb 23. PMID 36786515

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Patients: Subjects indicated for the treatment of AF with the cryoablation system according to current and future Guidelines and system indications for use
  Boston Scientific Cardiac Cryoablation System: cryoablation of atrial fibrillation consisting in electrical isolation of the pulmonary veins
  The enrolled patients will further be divided into:
  1. Treatment subjects (Followed for 12 months)
  2. Attempt subjects (study device inserted but not ablation treatment received)
  3. Intent subjects (study device not inserted)
  4. Consent ineligible (no meeting eligibility criteria after enrollment)
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 400
Completed | 359
Not Completed | 41
Not completed — Treatment - withdrawal by subject | 14
Not completed — Treatment - Lost to Follow-up | 11
Not completed — Treatment - End of study due to logistical reasons | 2
Not completed — Treatment - End of study due to refusing testing COVID | 1
Not completed — Treatment - Death | 1
Not completed — Treatment - Withdrawn due to unknown reason | 2
Not completed — Consent Ineligible - Does not meet eligibility criteria | 1
Not completed — Attempt | 2
Not completed — Intent | 7

BASELINE CHARACTERISTICS:
Population: Includes all treatment, attempt and intent subjects.
  Excludes Consent Ineligible patient and one attempt subject who, at the time of study withdrawal also withdrew their consent to have data included in future analyses.
Groups:
- Enrolled Patients: Subjects indicated for the treatment of AF with the cryoablation system according to current and future Guidelines and system indications for use
  Boston Scientific Cardiac Cryoablation System: cryoablation of atrial fibrillation consisting in electrical isolation of the pulmonary veins
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 251
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Black | 1
  Race: White | 256
  Race: Not Disclosed | 140
Region of Enrollment [Number; unit: participants]
  Netherlands | 47
  Belgium | 30
  Italy | 45
  United Kingdom | 54
  France | 109
  Germany | 105
  Croatia | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety Event Free Rate
Description: Freedom from procedure or device related adverse events after intervention, analyzed in all treatment and attempt subjects. The Primary Safety Endpoint is analyzed using data from all TREATMENT and ATTEMPT subjects including those with missing data. Subjects with missing data are censored at the appropriate timepoint in the KM analysis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Primary Safety Endpoint: The Primary Safety Endpoint is analyzed using data from all TREATMENT and ATTEMPT subjects.
Arm/Group | Primary Safety Endpoint
Number analyzed (Participants) | 391
Participants | 373

2. Primary Outcome: Failure Free Rate
Description: includes freedom from failure of intervention or more than one repeated procedures within 90 days post index procedure, or documented atrial fibrillation, new onset atrial flutter or atrial tachycardia between 91 days and 365 days post procedure
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Patients (Primary Effectiveness Endpoint): The Primary Effectiveness Endpoint is analyzed using data from all eligible TREATMENT subjects. Eligible TREATMENT subjects for the primary effectiveness endpoint includes all TREATMENT subjects who do not have an implantable continuous ECG recording system (eg. Pacemaker, arrhythmia loop recording systems, ICD, CRT).
Arm/Group | Treatment Patients (Primary Effectiveness Endpoint)
Number analyzed (Participants) | 355
Participants | 223

3. Secondary Outcome: Documentation and Rate of Acute Procedural Success
Description: Electrical isolation of a pulmonary vein (PV) is demonstrated at minimum by entrance block using the Cryo Mapping Catheter. The Secondary Effectiveness Endpoint is analyzed using data from all TREATMENT subjects.
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Groups:
- TREATMENT Patients (Secondary Effectiveness Endpoint): All Treatment patients
Arm/Group | TREATMENT Patients (Secondary Effectiveness Endpoint)
Number analyzed (Participants) | 390
Participants | 359

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 1/399
Serious Adverse Events (participants affected / at risk) | 71/399
Other Adverse Events (participants affected / at risk) | 47/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Patients (N=399)
3rd degree AV block (Cardiac disorders) | 1 (1)
Angina/Chest pain (Injury, poisoning and procedural complications) | 1 (1)
Atrial Fibrillation (AF) (Cardiac disorders) | 17 (18) — Including Atrial Fibrillation (AF) paroxysmal, AF persistent, AF recurrence, Atrial Tachycardia, hospital admission for AF
Implantation LBB Pacemaker (Cardiac disorders) | 1 (1)
Atrial Flutter (AFl) (Cardiac disorders) | 4 (5) — Including palpitations and hospital admissions
Atrial tachycardia/Other supraventricular tachycardia (Cardiac disorders) | 2 (2) — AV-nodal re-entry tachycardia (AVNRT), supraventricular tachycardia
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) — Intestine Cancer, Lobectomy, Suspicion of a carcinoid in the intestine, uterus cancer surgery and whipple/ (Endoscopic retrograde cholangiopancreatography) ERCP
CerebroVascular Accident (CVA) (Vascular disorders) | 2 (2) — benign paroxysmal position dizziness, ischemia
Chest Pain (General disorders) | 2 (2) — Chest pain, instable angina pectoris
Coronary Artery Disease (Vascular disorders) | 4 (4) — Coronary angiographia; electiv Recanalisation, actually without symptoms; Exclusion progress Coronary Artery Disease (CAD); Left main coronary artery intrastent restenosis
Dizziness (General disorders) | 1 (1) — domestic fall in benign positional vertigo
Dyspnea - Heart Failure (Cardiac disorders) | 1 (1) — Hisbundel Ablation
Embolism - Air (Injury, poisoning and procedural complications) | 1 (1) — ST elevation during ablation procedure.
Endocrine (Endocrine disorders) | 2 (2) — Hyperthyroid struma multinodosa both sides; Parathyroidectomie
COVID19 infection (Infections and infestations) | 1 (1)
Fistula (Aterial/Venous) (Injury, poisoning and procedural complications) | 3 (4) — Arteriovenous fistula; Fistula; Pain on the right femoral fistula; Right femoral arterio-venous fistula with hematoma
Gastritis (Injury, poisoning and procedural complications) | 1 (1) — Dyspnoe
Gastrointestinal (Gastrointestinal disorders) | 4 (4) — abdominal abces; Abdominal pain right lower abdomen; ileus, hernia umbilicalis; suspected appendicitis
Genitourinary (Renal and urinary disorders) | 1 (1) — urinary bladder tumor resection
Head, Eyes, Ears, Nose, Throat (HEENT) (General disorders) | 2 (3) — Cholesteatom right; nervus opticus inflammation;
Heart Failure symptoms - Unspecified (Cardiac disorders) | 2 (2) — CRT-D (cardiac resynchronization therapy - defibrillator) implant; worsening heart failure
Hematological (Blood and lymphatic system disorders) | 1 (1) — Anemia
Hematoma (Injury, poisoning and procedural complications) | 3 (3) — IHematoma, hematoma inguinal area, subcutaneous hematoma
Hypertension/Hypertensive Crisis (Vascular disorders) | 2 (2) — Hypertensive derailement
Integumentary (Skin and subcutaneous tissue disorders) | 2 (2) — Fever, melanoma of the skin
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) — carpal tunnel syndrom
Myocardial Infarction (Injury, poisoning and procedural complications) | 1 (1) — Post interventional STEMI (ST segment elevation myocardial infarction)
Myocardial perforation with tamponade (Injury, poisoning and procedural complications) | 2 (2) — drained tamponade, pericardial effusion
non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1) — ICD (implantable cardioverter defibrillator) Shock
Oozing/Bleeding (Injury, poisoning and procedural complications) | 2 (2) — Bleeding; Groin access site hematoma
Non Cardiovascular Pain (Injury, poisoning and procedural complications) | 1 (1) — chest pain due to gastric problems
Pericardial effusion (Injury, poisoning and procedural complications) | 1 (1) — right ventricular effusion
Phrenic nerve injury temporary (Injury, poisoning and procedural complications) | 1 (1)
Physical trauma (General disorders) | 4 (5) — Hand Fracture; Fracture of the neck and femur; right upper and lower limb motor deficit; spinal fracture following trauma; wound dehiscence
Procedure related Allergic reactions/Adverse drug reaction (Injury, poisoning and procedural complications) | 2 (2) — Bradycardy, Dizziness; Bronchospasm
Procedure related Pulmonary (including cough, hemoptysis) (Injury, poisoning and procedural complications) | 1 (1) — Hospital admission with AF,heamoptysis and fever
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (3) — acute dyspnea; Pneumonia with exacerbated COPD (Chronic Obstructive Pulmonary Disease); pneumopathy
Left renal colic (Renal and urinary disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stroke (Injury, poisoning and procedural complications) | 1 (1) — cerebellar infarctation left
Syncope (General disorders) | 1 (1)
Thrombus (Injury, poisoning and procedural complications) | 1 (1) — Femoral vein thrombosis
Transient Ischemic Attack (TIA) (Injury, poisoning and procedural complications) | 1 (1)
Pectoralis twitching due to pacemaker (Injury, poisoning and procedural complications) | 1 (1)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 1 (1)
Vessel trauma (Injury, poisoning and procedural complications) | 1 (1) — hematic leakage from collateral femoral artery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Patients (N=399)
Angina/Chest pain (Injury, poisoning and procedural complications) | 2 (2) — atypic thorax pain; Dyspnoe d'effort
Atrial Fibrillation (AF) (Cardiac disorders) | 4 (4) — Atrial fibrillation (AF); Hospital admission with AF; repeat ablation procedure
Atrial flutter (Cardiac disorders) | 3 (3) — tachycardia-like palpitations; Atrial flutter; Atypical Atrial flutter
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1)
Dyspnea - Heart Failure (Cardiac disorders) | 1 (1)
Embolism - Air (Injury, poisoning and procedural complications) | 1 (1)
Gastritis (Injury, poisoning and procedural complications) | 2 (2) — stomach ache; GERD (Gastroesophageal reflux disease) exacerbation
Gastroparesis (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 6 (6)
Hoarse Voice (Injury, poisoning and procedural complications) | 1 (1)
Oozing/Bleeding (Injury, poisoning and procedural complications) | 3 (3)
Pain (Non-cardiovascular) (Injury, poisoning and procedural complications) | 1 (1)
Pain cardiovascular (Non-ischemic) (Injury, poisoning and procedural complications) | 1 (1)
Pericarditis (Injury, poisoning and procedural complications) | 1 (1)
Phrenic nerve injury permanent (Injury, poisoning and procedural complications) | 1 (1)
Phrenic nerve injury temporary (Injury, poisoning and procedural complications) | 7 (7)
Procedure related Allergic reactions/Adverse drug reaction (Injury, poisoning and procedural complications) | 2 (2)
Procedure related Anesthesia/Sedation (Injury, poisoning and procedural complications) | 1 (1) — Keratitis
Procedure related Gastrointestinal (Injury, poisoning and procedural complications) | 2 (2) — Abdominal pain
Procedure related Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedure related Neurological (Non-TIA, non-stroke, dysphagia, speech disturbance/dysarthria) (Injury, poisoning and procedural complications) | 3 (3) — visual disturbance; migraine
Procedure related Pulmonary (including cough, hemoptysis) (Injury, poisoning and procedural complications) | 3 (3) — Dyspnoe, hemoptysis
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Psychological issues related to Phrenic Nerve Injury (PNI) (Injury, poisoning and procedural complications) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Visual blurring/Disturbances (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04250714/Prot_SAP_000.pdf